CLINICAL TRIAL: NCT00846092
Title: Phase 1 Study To Determine the Effects of Short Term Near-infrared Light (NIR) Therapy on Anatomic and Functional Abnormalities of Diabetic Macular Edema, and Assess Safety of Short Term Near-infrared Light Therapy in Eyes With Diabetic Macular Edema.
Brief Title: Near-infrared Light (NIR) Therapy for Diabetic Macular Edema: A Pilot Study
Acronym: NIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: The New York Eye & Ear Infirmary (Other)
Responsible Party: Principal Investigator, Harry T Whelan, MD, PI, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIR for Diabetic Maculopathy
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Retinopathy; Diabetic Macular Edema; NIR; Near-infrared Light Therapy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental): * The study will require 20 subjects.
  * Each subject will have one "study eye" that will be designated for treatment.
  * Subjects will be exposed to light emitted from Warp 10 LED's (Quantum Devices, Barneveld, WI) at wavelengths of 670 nm (+/-15nm) with a minimum exposure of 4 J/cm2 (4.0 - 7.68J/cm2). This is accomplished by applying the 50 mW/cm2 (50 - 80 mw/cm2) LED-generated light to the study eye.
  * Treatments involve application of the LED-generated light for 80 seconds, twice daily.
  Primary efficacy and toxicity outcomes are determined by measuring excess retinal thickness via Ocular Coherence Tomography at 1 month, 3 months, and 6 months, prior to conclusion of the study.
  • This protocol will be stopped if, at any point in the study, a 50% increase in excess retinal thickness is demonstrated via OCT in 25% of subjects in the experimental group.
  Interventions: Device: Warp 10 LED Device; Device: Near-infrared light (NIR)

INTERVENTIONS:
Device: Warp 10 LED Device — Study Subjects will take the Warp 10 (LED) home and treat twice per day for three months
  Other Names: Warp 10
Device: Near-infrared light (NIR) — * Subjects will be exposed to light emitted from LED's at wavelengths of 670 nm (+/-15nm) with a minimum exposure of 4 J/cm2 (4.0 - 7.68J/cm2). This is accomplished by applying the 50 mW/cm2 (50 - 80 mw/cm2) LED-generated light to the study eye.
  * Treatments involve application of the LED-generated light for 80 seconds, twice daily.
  Other Names: Warp 10 LED's

SUMMARY:
Summary of Study Rationale Near-infrared light (NIR) via light-emitting diodes (LED) treatment promotes retinal healing and improve visual function following high intensity laser retinal injury by augmenting cellular energy metabolism, enhances mitochondrial function, increases cytochrome C oxidase activity, stimulates antioxidant protective pathways, and promotes cell survival. LED directly benefits injured neurons in the retina, the lateral geniculate nucleus, and the visual cortex, where perception occurs. From a public health perspective, a Light-Emitting Diode (LED) Array study is important to conduct because it has been approved as a non-significant risk (NSR) device for treatment of eye disorders, it has a low cost of treatment, and it may serve as an effective, non-invasive alternative or adjunctive treatment to laser photocoagulation, the current standard of care for DME.

Study Objectives and Hypotheses

1. To determine the effects of short term (3 month) near-infrared light (NIR) therapy on anatomic and functional abnormalities of diabetic macular edema as assessed by visual acuity, optical coherence tomography, multifocal electroretinography (mERG) and fundus bimicroscopy.
2. To assess safety of short term near-infrared light therapy in eyes with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years Subjects <18 years old are not being included because DME is so rare in this age group that the diagnosis of DME may be questionable.
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   • Any one of the following will be considered to be sufficient evidence that diabetes is present: Current regular use of insulin for the treatment of diabetes Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes Documented diabetes by ADA and/or WHO criteria (see Procedures Manual for definitions)
3. At least one eye meets the study eye criteria.
4. Fellow eye meets criteria.
5. Able and willing to provide informed consent.
6. Any candidate identified by a study investigator as being able to successfully tolerate a 3 month deferral of laser photocoagulation.

   Exclusion Criteria:
7. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
8. Subjects in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
9. Participation in an investigational trial within 30 days of NIR participation that involved treatment with any drug that has not received regulatory approval at the time of study entry.

   • Note: subjects cannot receive another investigational drug while participating in the study during the first 6 months...
10. Major surgery within 28 days prior to participation or major surgery planned during the next 6 months.

    • Major surgery is defined as a surgical procedure that is more extensive than fine needle biopsy/aspiration, placement of a central venous access device, removal/biopsy of a skin lesion, or placement of a peripheral venous catheter.
11. Subject is expecting to move out of the area during the 6 months of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Excess retinal thickness on OCT at 1 month, 3 months and 6 months. goal = reduce excess thickness by at least 50% | 1 month, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harry T Whelan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Moss SE, Klein R, Klein BE. Ten-year incidence of visual loss in a diabetic population. Ophthalmology. 1994 Jun;101(6):1061-70. doi: 10.1016/s0161-6420(94)31217-6. PMID 8008348
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group; Lachin JM, Genuth S, Cleary P, Davis MD, Nathan DM. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive therapy. N Engl J Med. 2000 Feb 10;342(6):381-9. doi: 10.1056/NEJM200002103420603. PMID 10666428
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Beauvoit B, Kitai T, Chance B. Contribution of the mitochondrial compartment to the optical properties of the rat liver: a theoretical and practical approach. Biophys J. 1994 Dec;67(6):2501-10. doi: 10.1016/S0006-3495(94)80740-4. PMID 7696489
- [Background] Karu T. Primary and secondary mechanisms of action of visible to near-IR radiation on cells. J Photochem Photobiol B. 1999 Mar;49(1):1-17. doi: 10.1016/S1011-1344(98)00219-X. PMID 10365442
- [Background] Wong-Riley MT, Liang HL, Eells JT, Chance B, Henry MM, Buchmann E, Kane M, Whelan HT. Photobiomodulation directly benefits primary neurons functionally inactivated by toxins: role of cytochrome c oxidase. J Biol Chem. 2005 Feb 11;280(6):4761-71. doi: 10.1074/jbc.M409650200. Epub 2004 Nov 22. PMID 15557336
- [Background] Liang HL, Whelan HT, Eells JT, Meng H, Buchmann E, Lerch-Gaggl A, Wong-Riley M. Photobiomodulation partially rescues visual cortical neurons from cyanide-induced apoptosis. Neuroscience. 2006 May 12;139(2):639-49. doi: 10.1016/j.neuroscience.2005.12.047. Epub 2006 Feb 7. PMID 16464535
- [Background] Eells JT, Wong-Riley MT, VerHoeve J, Henry M, Buchman EV, Kane MP, Gould LJ, Das R, Jett M, Hodgson BD, Margolis D, Whelan HT. Mitochondrial signal transduction in accelerated wound and retinal healing by near-infrared light therapy. Mitochondrion. 2004 Sep;4(5-6):559-67. doi: 10.1016/j.mito.2004.07.033. PMID 16120414
- [Background] Whelan HT, Connelly JF, Hodgson BD, Barbeau L, Post AC, Bullard G, Buchmann EV, Kane M, Whelan NT, Warwick A, Margolis D. NASA light-emitting diodes for the prevention of oral mucositis in pediatric bone marrow transplant patients. J Clin Laser Med Surg. 2002 Dec;20(6):319-24. doi: 10.1089/104454702320901107. PMID 12513918
- [Background] Whelan HT, Buchmann EV, Dhokalia A, Kane MP, Whelan NT, Wong-Riley MT, Eells JT, Gould LJ, Hammamieh R, Das R, Jett M. Effect of NASA light-emitting diode irradiation on molecular changes for wound healing in diabetic mice. J Clin Laser Med Surg. 2003 Apr;21(2):67-74. doi: 10.1089/104454703765035484. PMID 12737646
- [Background] Wong-Riley MT, Bai X, Buchmann E, Whelan HT. Light-emitting diode treatment reverses the effect of TTX on cytochrome oxidase in neurons. Neuroreport. 2001 Oct 8;12(14):3033-7. doi: 10.1097/00001756-200110080-00011. PMID 11568632
- [Background] Eells JT, Henry MM, Summerfelt P, Wong-Riley MT, Buchmann EV, Kane M, Whelan NT, Whelan HT. Therapeutic photobiomodulation for methanol-induced retinal toxicity. Proc Natl Acad Sci U S A. 2003 Mar 18;100(6):3439-44. doi: 10.1073/pnas.0534746100. Epub 2003 Mar 7. PMID 12626762
- [Background] Kowluru RA, Atasi L, Ho YS. Role of mitochondrial superoxide dismutase in the development of diabetic retinopathy. Invest Ophthalmol Vis Sci. 2006 Apr;47(4):1594-9. doi: 10.1167/iovs.05-1276. PMID 16565397
- [Background] Kowluru RA, Kowluru V, Xiong Y, Ho YS. Overexpression of mitochondrial superoxide dismutase in mice protects the retina from diabetes-induced oxidative stress. Free Radic Biol Med. 2006 Oct 15;41(8):1191-6. doi: 10.1016/j.freeradbiomed.2006.01.012. Epub 2006 Feb 6. PMID 17015165
- [Background] Nyengaard JR, Ido Y, Kilo C, Williamson JR. Interactions between hyperglycemia and hypoxia: implications for diabetic retinopathy. Diabetes. 2004 Nov;53(11):2931-8. doi: 10.2337/diabetes.53.11.2931. PMID 15504974
- [Background] Obrosova IG, Stevens MJ, Lang HJ. Diabetes-induced changes in retinal NAD-redox status: pharmacological modulation and implications for pathogenesis of diabetic retinopathy. Pharmacology. 2001;62(3):172-80. doi: 10.1159/000056091. PMID 11287819
- [Background] Weinberger D, Axer-Siegel R, Landau D, Yassur Y. Retinal thickness variation in the diabetic patient measured by the retinal thickness analyser. Br J Ophthalmol. 1998 Sep;82(9):1003-6. doi: 10.1136/bjo.82.9.1003. PMID 9893588